CLINICAL TRIAL: NCT06805526
Title: Does Intermittent Islamic Fasting Have Beneficial Effect in Management of Metabolic Syndrome? a Randomized Control Trial
Brief Title: Role of Intermittent Islamic Fasting in Management of Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hanaa Abu Elazayem Ibrahim Nofal, Principal Investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Intermittent Islamic fasting
Record Dates: First submitted 2025-01-22; First posted 2025-02-03 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Intermittent Islamic Fasting in Metabolic Syndrome
Keywords: Intermittent Islamic Fasting, lifestyle modification and Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: At first, a Sample was picked by systematic random technique from patients attending clinical nutrition outpatient clinic of Zagazig University hospital then by block randomization, according to sex and BMI, the sample was classified randomly according to intervention type by block randomization using sealed Envelope website into 6 blocks each block size 9 list length with allocation ratio 1:1, Study was open -label . The sample was divided into two groups (intervention group and control group).
Masking Description: None (open label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Active Comparator): follow Islamic fasting with lifestyle modification
  Interventions: Behavioral: Intermittent Islamic fasting with lifestyle modification
- Control group (Sham Comparator): follow lifestyle modification only
  Interventions: Behavioral: Lifestyle modification only

INTERVENTIONS:
Behavioral: Intermittent Islamic fasting with lifestyle modification — Both groups followed a healthy lifestyle for 6 months including:
  Diet: The participants' habitual total energy expenditure was estimated using the standard Harris-Benedict equation. To achieve a reduction of over 500 kcal/day, a daily intake of 1,200 to 1,500 kcal is typically recommended for women and 1,500 to 1,800 kcal for men .
  Physical Activity: Moderate physical activity is advised. This includes engaging in exercise for 30 to 60 minutes, five days a week. Additionally, incorporating resistance training is recommended twice a week .
  * stress management How to cope with stress, relaxation technique, quality and quantity of sleep,
  * Drinking enough water 30-40ml/kg/day. Followed Intermittent Islamic fasting which meant fasting two days per week (Monday and Thursday) with fasting (13, 14, 15) middle of lunar months. (during Intermittent Islamic fasting caloric requirement was distributed as 30-40
  For Group I (intervention group) only, Followed Intermittent Islamic fasting wh
  Arms: Intervention group
Behavioral: Lifestyle modification only — The participants' habitual total energy expenditure was estimated using the standard Harris-Benedict equation. For men, the formula is: BMR = 66.4730 + 13.7516 × weight (kg) + 5.0033 × height (cm) - 6.7550 × age (years). For women, the formula is: BMR = 655.0955 + 9.5634 × weight (kg) + 1.8496 × height (cm) - 4.6756 × age (years) [27]. To achieve a reduction of over 500 kcal/day, a daily intake of 1,200 to 1,500 kcal is typically recommended for women and 1,500 to 1,800 kcal for men [28].
  Physical Activity: Moderate physical activity is advised. This includes engaging in exercise for 30 to 60 minutes, five days a week. Additionally, incorporating resistance training is recommended twice a week [29].
  * stress management How to cope with stress, relaxation technique, quality and quantity of sleep,
  * Drinking enough water 30-40ml/kg/day.
  Arms: Control group

SUMMARY:
Metabolic syndrome doubles the risk of developing cardiovascular diseases and type 2 diabetes mellitus. Intermittent Islamic fasting is an effective health strategy associated with various benefits. Objectives: to compare effect of Intermittent Islamic fasting with lifestyle modification versus lifestyle modification only on weight management, blood pressure, blood glucose and lipid profile among a group of metabolic syndrome patients.

DETAILED DESCRIPTION:
Metabolic Syndrome (MetS), also called "Syndrome X" or "insulin resistance syndrome," describes a common condition characterized by high blood pressure, elevated triglycerides, central obesity, and low HDL cholesterol levels . Having metabolic syndrome doubles the risk of developing cardiovascular diseases and type 2 diabetes mellitus. The prevalence of Metabolic Syndrome (MetS) is globally increasing due to the widespread adoption of the Western lifestyle . Between 2011 and 2018, the prevalence of Metabolic Syndrome (MetS) in the USA significantly increased from 37.6% in 2011-2012 to 41.8% in 2017-2018. This trend may be indicative of the rising epidemic of type 2 diabetes there . In Egypt, an estimated 10.9 million people currently have diabetes. This number is projected to rise to 13 million by 2030 and to 20 million by 2045.our aim to compare effect of Intermittent Islamic fasting with lifestyle modification versus lifestyle modification only on weight management, blood pressure, blood glucose and lipid profile among a group of metabolic syndrome patients.

A Randomized control open label trial was conducted on with metabolic syndrome, their ages range from (30- 45 years) attending the clinical nutrition outpatient clinic in the Zagazig University hospital from 1st of August (2023) to the end of February (2024) using consort guidelines and flow chart were used in this study including 54 patients with metabolic syndrome. At first, a Sample was picked by systematic random technique from patients attending clinical nutrition outpatient clinic of Zagazig University hospital then by block randomization, according to sex and BMI, the sample was classified randomly according to intervention type by block randomization using sealed Envelope website into 6 blocks each block size 9 list length with allocation ratio 1:1, Study was open -label . The sample was divided into two groups (intervention group and control group).

1. Group I: intervention group (27 patients) followed Islamic fasting with lifestyle modification; (Islamic fasting means: fasting two days per week (Monday and Thursday) with fasting (13, 14, 15) middle of lunar months).
2. Group II: control group (27 patients) followed lifestyle modification only.

ELIGIBILITY:
Inclusion Criteria:

* Adults with metabolic syndrome
* Adults (30-45years old)
* providing a consent.

Exclusion Criteria:

* Had any chronic diseases
* pregnant females.

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Changes in Body weight | 6 months
  Pre and Post measurements of body weight in kilograms
Change in waist circumference | 6 months
  Pre and Post measurements of waist circumference in centimeters
Changes in Body mass index | 6 months
  Pre and Post measurements of Body mass index in kg/m^2
Changes in blood pressure | 6 months
  Periodic measurements in systolic and diastolic blood pressure in mmHg

SECONDARY OUTCOMES:
Lipid profile Assessment | 6 months
  pre and post intervention measurements of serum Triglycerides, cholesterol, High density lipoprotein and Low density lipoprotein levels
Fasting blood glucose level | 6 months
  Pre and post intervention measurements of fasting blood glucose level

CONTACTS AND LOCATIONS:
Overall Officials: Hanaa A Nofal, MD, Principal Investigator — Zagazig University
Locations (1):
- Zagazig University outpatients clinics, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nofal HA, Elmor AAR, AbdAllah AM, Zaitoun NA, Andargeery SY, Sharafeddin MA, Hassan RIA, Elhawy LL. Effect of intermittent Islamic fasting in management of metabolic syndrome: a randomized control trial. BMC Public Health. 2025 Jul 16;25(1):2476. doi: 10.1186/s12889-025-23493-7. PMID 40670993